CLINICAL TRIAL: NCT02430545
Title: A Phase 1, Open-label, Fixed-sequence, 2-period Study In Healthy Volunteers To Investigate The Effect Of Multiple Doses Of Rifampin On Single Dose Glasdegib (Pf-04449913) Plasma Pharmacokinetics
Brief Title: Understanding The Effect Of A Strong CYP3A4 Inducer On Glasdegib Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1371015
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Volunteers
Keywords: Glasdegib; PF-04449913; Drug-drug interaction; CYP3A4 inducer; Pharmacokinetics
MeSH Terms: interventions — glasdegib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glasdegib, Rifampin (Experimental): Subjects receive a 100mg oral dose of glasdegib under fasted conditions with washout, then single 100mg oral dose of glasdegib under fasted following dosing to steady state with rifampin
  Interventions: Drug: Glasdegib; Drug: Rifampin

INTERVENTIONS:
Drug: Glasdegib — Subjects receive a 100mg oral dose of glasdegib under fasted conditions with washout, then single 100mg oral dose of glasdegib under fasted following dosing to steady state with rifampin
Drug: Rifampin — Subjects receive rifampin 600 mg oral dose daily [Day -6 to day 4]

SUMMARY:
The study also aims to determine the effect of a strong enzyme (CYP3A4) inducer-rifampin- on drug exposure of Glasdegib. This study will be conducted in healthy subjects given a single dose of glasdegib in each period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Female subjects of non childbearing potential must meet at least one of the following criteria:

  1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; AND have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure.
* All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* A positive urine drug screen
* Screening supine 12 lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Subjects with family history of myocardial infarction, congenital long QT syndrome, torsades de pointes or clinically significant ventricular arrhythmias.
* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use two highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product and, refrain from sperm donation for the duration of the study and for at least 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 5 days
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 5 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 5 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Apparent Oral Clearance (CL/F) | 5 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 5 days
Apparent Volume of Distribution (Vz/F) | 5 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 5 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Shaik MN, Hee B, Wei H, LaBadie RR. Evaluation of the effect of rifampin on the pharmacokinetics of the Smoothened inhibitor glasdegib in healthy volunteers. Br J Clin Pharmacol. 2018 Jun;84(6):1346-1353. doi: 10.1111/bcp.13568. Epub 2018 Apr 10. PMID 29488303